CLINICAL TRIAL: NCT00630175
Title: Evaluation of the Hypnotic Properties of Zolpidem-MR 12.5 mg and Zolpidem 10 mg Marketed Product Compared to Placebo in Patients With Primary Insomnia. A Double-Blind, Randomized, Placebo-Controlled,Three Way Cross-Over Study
Brief Title: Evaluation of the Hypnotic Properties of Zolpidem-MR 12.5 mg and Zolpidem 10 mg Marketed Product Compared to Placebo in Patients With Primary Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5202
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: zolpidem-MR (modified release)
Drug: zolpidem (SL800750)
Drug: placebo

SUMMARY:
The primary objective is to evaluate the hypnotic efficacy of zolpidem-MR (modified release) 12.5 mg and zolpidem 10 mg marketed product in comparison with placebo in patients with primary insomnia and sleep maintenance difficulties, using polysomnography (PSG) recordings and patient sleep questionnaires.

The secondary objective is to evaluate the clinical safety and tolerability of zolpidem-MR 12.5 mg and zolpidem 10 mg marketed product in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia based on Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2003-09; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Polysommography (PSG) wake time after sleep onset (WASO)

SECONDARY OUTCOMES:
PSG parameters, Patient's sleep questionnaire, Patient's global impression, Relative degree of satisfaction with the different study drugs

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Laval, Canada